CLINICAL TRIAL: NCT03921606
Title: Using Information Communication Technology (Whatsapp/WeChat) to Deliver Brief Motivational Interviewing (i-BMI) to Promote Smoking Cessation Among Smokers With Chronic Diseases
Brief Title: Using ICT to Deliver Brief Motivational Interviewing to Promote Smoking Cessation Among Smokers With Chronic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NTWCREC19001
Record Dates: First submitted 2019-03-04; First posted 2019-04-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive a brief MI via WhatsApp/WeChat on a smartphone during the study period. The brief MI messages will be delivered more intensively as preferred by the subject (usually not less than once every 2 to 3 days and no more than 2 times per day) for the first 6 months. The frequency of delivering the messages via WhatsApp/WeChat will be interactive, depending on the subjects' actions and responses, and may take several sessions of chats within several days or weeks. However, the total time spent by the interventionist will not be more than that for a traditional MI with several long sessions. After 6 months, minimal messages will be provided to the subjects by merely following their progress of behavioural changes and responding to their questions to maintain contact until the 1-year follow-up. The total time spent will be recorded and analysed.
  Interventions: Behavioral: Motivational Interviewing (i-BMI)
- Control group (Other): The control group will receive individual face-to-face generic health advice (about 5 minutes) on a health-related lifestyle practice such as eating more vegetables and fruits, eating less high salt, fat or sugar foods, consuming less sugary drinks, engaging in more exercise of any kind or intensity, reducing alcohol consumption or reducing weight (if overweight or obese) in SOPCs. A self-help booklet on smoking cessation published by the Hong Kong Council on Smoking and Health with Hotline will be also provided in the SOPCs. The subjects in this group will receive the same schedule of follow-ups as in the intervention group, but they will not receive any follow-up booster intervention.
  Interventions: Behavioral: Individual face-to-face generic health advice

INTERVENTIONS:
Behavioral: Motivational Interviewing (i-BMI) — A brief MI via WhatsApp/WeChat
  Arms: Experimental group
Behavioral: Individual face-to-face generic health advice — Individual face-to-face generic health advice (about 5 minutes) on a health-related lifestyle practice such as eating more vegetables and fruits, eating less high salt, fat or sugar foods, consuming less sugary drinks, engaging in more exercise of any kind or intensity, reducing alcohol consumption or reducing weight (if overweight or obese). A self-help booklet on smoking cessation published by the Hong Kong Council on Smoking and Health with Hotline will be also provided in the SOPCs.
  Arms: Control group

SUMMARY:
This study aims to evaluate the effectiveness of a general health promotion (GHP) approach using information communication technology (ICT) to deliver a brief motivational interviewing (MI) to motivate smokers with chronic diseases to quit smoking. Subjects in the intervention group will receive a GHP approach using ICT (e.g., WhatsApp/WeChat) to deliver brief MI. Subjects in the control group will receive an individual face-to-face generic health advice plus a self-help booklet on smoking cessation at the time of recruitment.

DETAILED DESCRIPTION:
Smoking exerts harmful effects on nearly every organ of the body and causes 7 million deaths worldwide each year. In Hong Kong, despite a decrease in the prevalence of daily cigarette smoking from 23.3% in 1982 to 10.0% in 2017, there are still 615,000 daily smokers. The evidence has shown that continued smoking in patients with chronic diseases can reduce the efﬁcacy of medical treatments and increase the risk of treatment-related side effects. Nevertheless, many smokers with chronic diseases have a long smoking history, a strong nicotine dependency, and have not attempted or have no intention to quit. It is essential to develop and evaluate a more innovative and effective intervention to enhance the acceptability of smoking cessation for smokers with chronic diseases.

The proposed intervention will aim to facilitate the movement through five stages of change (pre-contemplation, contemplation, preparation, action and maintenance)15 via the (i) foot-in-the-door technique and (ii) a brief MI. The World Health Organization defines medical and public health practice supported by mobile devices as mobile health, a new strategy to promote health.21 Instant messaging, such as WhatsApp/WeChat delivered by mobile devices, is widely used for health promotion and treatment compliance.22 One advantage of using WhatsApp/WeChat is that it can offer quick, real-time interactions and continuing professional advice and support for subjects to manage their health-related lifestyle practices. Most importantly, WhatsApp/WeChat is more flexible, efficient and time-saving compared to face-to-face meetings to deliver a brief MI as face-to-face meetings would require the subjects to return several times for interventions. A systematic review of the use of mobile phone-based interventions for smoking cessation showed that smokers who received instant messages via mobile phones were more likely to abstain from smoking compared to those who used traditional face-to-face cessation services.23 A recent study conducted by our team in Hong Kong also showed that the use of WhatsApp for instant messaging was more effective in smoking relapse prevention for recent quitters.24 However, we found no reports or proposals based on the above conceptual framework and strategies in which ICTs were used with smokers who had no intention to quit.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above,
* able to speak Cantonese and read Chinese
* do not intend to quit smoking (pre-contemplation stage), but are willing to promote their health
* use a smartphone and can use an instant messaging tool (e.g., WhatsApp/WeChat)
* willing to receive health promotion advice and interact with our interventionist via WhatsApp/WeChat on a smartphone throughout the study period

Exclusion Criteria:

* inability to give informed consent or participate in our intervention due to impaired mental status, cognitive impairment or communication barriers
* participate in another smoking cessation programme or service

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence at 6 months | 6-month follow-up
  The biochemically validated smoking abstinence will be confirmed by a saliva cotinine level of less than 115 ng/ml in parallel test and a carbon monoxide level in expired air of less than 9 parts per million (ppm)

SECONDARY OUTCOMES:
biochemically validated smoking abstinence at 12 months | 12-month follow-up
  The biochemically validated smoking abstinence will be confirmed by a saliva cotinine level of less than 115 ng/ml in parallel test and a carbon monoxide level in expired air of less than 9 parts per million (ppm)
Self-reported 7-day point prevalence of smoking abstinence at 6 and 12 months | 6- and 12-month follow-up
  Structured questionnaires will be developed by adopting or modifying international and/or locally validated instruments.
Any behavioural change reported by the subjects at 3, 6 and 12 months | 3-, 6- and 12-month follow-ups
  EQ-5D five-level questionnaire (EQ-5D-5L) will be administered at 3, 6, and 12 months. Chinese-specific EQ-5D-5L value set will enable the estimation of EQ-5D-5L health utility scores applicable for Chinese population.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No